CLINICAL TRIAL: NCT04358666
Title: Evaluation of the Best Treatment in Terms of Quality of Life for Patients Having a Brain Metastasis
Acronym: OPTMETACER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 19-086
Record Dates: First submitted 2020-03-31; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-03

CONDITIONS: Quality of Life; Brain Metastases
Keywords: brain metastasis, best treatment, quality of life, surgery+radiosurgery, hypofractionned radiosurgery
MeSH Terms: conditions — Brain Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: randomization between surgery and focal radiosurgery of the surgical site and hypofractionned radiosurgery of the tumor
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery and focal radiosurgery of the surgical site (Active Comparator)
  Interventions: Procedure: surgery and focal radiosurgery of the surgical bed
- hypofractionned radiosurgery (Active Comparator)
  Interventions: Procedure: surgery and focal radiosurgery of the surgical bed

INTERVENTIONS:
Procedure: surgery and focal radiosurgery of the surgical bed — hypofractionned radiosurgery of the lesion
  Other Names: hypofractionned radiosurgery of the lesion

SUMMARY:
Main Goal : evaluation of quality of life for patient having a brain metastasis and allowed to have either surgery and radiosurgery of the surgical site or only hypofractionned radiosurgery on the lesion.

second objectives : evaluation of the local control of the disease evaluation of the overall survival interval without progression evaluation of the medico economic performance of each treatment protocol neuro cognitive evaluation at the end of the protocol

DETAILED DESCRIPTION:
A patient with a brain metastasis may have the choice between surgery and focal radiosurgery of the surgical site and only hypofractionned radiosurgery on the lesion.

No previous study has focused on quality of life regarding these two treatments options.

ELIGIBILITY:
Inclusion Criteria:

* eligible for both treatments options OMS status <3 primary cancer with no evolution brain metastasis < 3cm ou giving symtoms patient with informed consent patient affilated to french social security

Exclusion Criteria:

* OMS > 3 More than 3 brain metastasis brain metastasis already treated with hypofractionned radiosurgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03-06 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
quality of life EORTC QLQ C30 | change between baseline and 6 month
  score European Organisation for Research and Treatment of Cancer Quality Life Quotation C30

SECONDARY OUTCOMES:
local control of the desease | baseline up to 24 month
survival without progression | 24 month
overall survival | 24 month
medico economic evaluation | 24 month
  cost-utility analysis
neuro cognitive evaluation | 12 and 24 month
  BOSTON NAMING TEST

CONTACTS AND LOCATIONS:
Locations (1):
- CHU CAEN, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided